CLINICAL TRIAL: NCT03399929
Title: Effects of Rehabilitation Following Traumatic Brain Injury and Stroke: A Long Term Outcome Study.
Brief Title: Traumatic Brain Injury and Stroke Long Term Outcome
Status: Recruiting | Type: Observational
Sponsor: Centre for Neuro Skills (Industry)
Responsible Party: Sponsor
Other Study IDs: LTO1
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Traumatic Brain Injury; Stroke
Keywords: Rehabilitation; Long term outcome
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TBI + Rehabilitation: Traumatic Brain Injury patients that received post acute rehabilitation
  Interventions: Other: Post Acute Rehabiltation
- TBI + No Rehabilitation: Traumatic Brain Injury patients that did not receive post acute rehabilitation
- CVA + Rehabilitation: Stroke patients that received post acute rehabilitation
  Interventions: Other: Post Acute Rehabiltation
- CVA + No Rehabilitation: Stroke patients that did not received post acute rehabilitation

INTERVENTIONS:
Other: Post Acute Rehabiltation
  Groups: CVA + Rehabilitation; TBI + Rehabilitation

SUMMARY:
Investigators will determine the long-lasting effects of post-acute rehabilitation after traumatic brain injury and stroke. Investigators will also evaluate if the beneficial effects of rehabilitation continue after discharge from a rehabilitative program.

DETAILED DESCRIPTION:
The long-term effects of rehabilitation will be evaluated on 60 patients with traumatic brain injury (TBI) and 60 patients that suffered a cerebrovascular accident (CVA) that underwent an comprehensive rehabilitative. These patients will be matched with subjects that received limited or no rehabilitation rehabilitative therapy. Thus, the total number of subjects in this study will be 240. Subjects will be contacted at least 1 year after discharge and will be lowed up every two-years thereafter for a total period of 10 years. Procedures will be performed in-person whenever possible. However, it is highly likely that the majority of participants will be contacted via phone interviews.

Aim 1: Determine if rehabilitation improves vocational status and living status after TBI and CVA.

Aim 2: Determine if rehabilitation improves life quality after TBI and CVA.

Aim 3: Determine if rehabilitation improves cognitive function after TBI and CVA.

Aim 4: Determine if rehabilitative benefits are sustained.

Aim 5: Determine if long-term outcome is dependent on the duration of rehabilitation.

Aim 6: Determine if long-term outcome is dependent on the nature of the rehabilitative treatment by comparing the effects of different types of rehabilitation. These will include the following: residential-multidisciplinary, day-treatment (i.e. full time multidisciplinary outpatient), outpatient (part-time), skilled nursing and no post-acute rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Endured a traumatic brain injury or stroke
* Subject or caretaker should be Fluent in English

Exclusion Criteria:

* Diagnosis of degenerative neurological disease prior to sustaining stroke or traumatic brain injury
* b) A history of major psychosis as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-V) prior to sustaining stroke or traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with a traumatic brain injury or stroke
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-05-04 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2028-05-04 (Estimated)

PRIMARY OUTCOMES:
Effects of rehabilitation on long term occupational Status after injury | 1 to 10 years
  Occupational Status Questionnaire
Effects of rehabilitation on long term cognitive function after injury | 1 to 10 years
  Brief Test of Adult Cognition by Telephone
Effects of rehabilitation on long term disability function after injury | 1 to 10 years
  Supervision Rating Scale and Disability Rating Scale
Effects of rehabilitation on long term quality of life after injury | 1 to 10 years
  Quality of Life in Neurological Disorders Measures (NeuroQOL)

SECONDARY OUTCOMES:
Effects of rehabilitation on long term health after injury | 1 to 10 years
  TBI and Health in Adults Questionnaire

OTHER OUTCOMES:
Effects of rehabilitation on post mortem health after injury | 1 to 10 years
  Post- Mortem health Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Griesbach, PhD, Principal Investigator — Centre for Neuro Skills
Locations (1):
- Centre for Neuro Skills, Encino, California, United States

IPD SHARING:
Plan to Share IPD: Undecided